CLINICAL TRIAL: NCT06323928
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled, Dose-finding Trial of Lu AG09222 for the Prevention of Migraine in Participants With Unsuccessful Prior Preventive Treatments
Brief Title: A Dose-finding Trial With Lu-AG09222 in Adults With Migraine Who Have Not Been Helped by Prior Preventive Treatments
Acronym: PROCEED
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20297A; 2023-508821-28-00 (Other: EU Trial)
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Headache; Chronic Migraine; Episodic Migraine
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Group A: Placebo SC (closed for recruitment) (Placebo Comparator): Participants will receive 2 injections of placebo.
  Interventions: Drug: Placebo
- Group B: Lu AG09222 SC (closed for recruitment) (Experimental): Participants will receive 1 injection of placebo and 1 injection containing Lu AG09222.
  Interventions: Drug: Lu AG09222; Drug: Placebo
- Group C: Lu AG09222 SC (closed for recruitment) (Experimental): Participants will receive 1 injection of placebo and 1 injection containing Lu AG09222.
  Interventions: Drug: Lu AG09222; Drug: Placebo
- Group D: Lu AG09222 SC (closed for recruitment) (Experimental): Participants will receive 1 injection of placebo and 1 injection containing Lu AG09222.
  Interventions: Drug: Lu AG09222; Drug: Placebo
- Group E: Lu AG09222 SC (closed for recruitment) (Experimental): Participants will receive 2 injections, each containing Lu AG09222.
  Interventions: Drug: Lu AG09222
- Group F: Placebo IV (Placebo Comparator): Participants will receive placebo by intravenous (IV) infusion.
  Interventions: Drug: Placebo
- Group G: Lu AG09222 IV (Experimental): Participants will receive Lu AG09222 by IV infusion.
  Interventions: Drug: Lu AG09222
- Group H: Lu AG09222 IV (Experimental): Participants will receive Lu AG09222 by IV infusion.
  Interventions: Drug: Lu AG09222
- Group I: Lu AG09222 IV (Experimental): Participants will receive Lu AG09222 by IV infusion.
  Interventions: Drug: Lu AG09222

INTERVENTIONS:
Drug: Lu AG09222 — Lu AG09222 will be administered per the arm description.
  Arms: Group B: Lu AG09222 SC (closed for recruitment); Group C: Lu AG09222 SC (closed for recruitment); Group D: Lu AG09222 SC (closed for recruitment); Group E: Lu AG09222 SC (closed for recruitment); Group G: Lu AG09222 IV; Group H: Lu AG09222 IV; Group I: Lu AG09222 IV
Drug: Placebo — Placebo matching to Lu AG09222 will be administered per the arm description
  Arms: Group A: Placebo SC (closed for recruitment); Group B: Lu AG09222 SC (closed for recruitment); Group C: Lu AG09222 SC (closed for recruitment); Group D: Lu AG09222 SC (closed for recruitment); Group F: Placebo IV

SUMMARY:
The purpose of this trial is to determine which doses of Lu AG09222 are recommended to help prevent migraines. People who join this trial have already tried 1 to 4 other available medications to prevent their migraines, but these medications have not helped them.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has a diagnosis of migraine as defined by International Classification of Headache Disorders Third Edition (ICHD-3) guidelines confirmed at the Screening Visit.
* The participant has a history of migraine onset ≥ 12 months prior to the Screening Visit.
* The participant has a migraine onset at ≤50 years of age.
* The participant has ≥4 migraine days per month for each month within the past 3 months prior to the Screening Visit.
* The participant has documented evidence of treatment failure in the past 10 years of at least 1 to 4 (maximum) different migraine preventive medications.

Key Exclusion Criteria:

* The participant has previously been dosed with an anti-pituitary adenylate cyclase-activating peptide (anti-PACAP treatment).
* The participant has confounding and clinically significant pain syndromes.
* The participant has a diagnosis of acute or active temporomandibular disorder.
* The participant has a history or diagnosis of confounding headaches.

Additional protocol-defined criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 874 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Number of Monthly Migraine Days (MMDs) | Baseline up to Week 12 (Weeks 1-12)

SECONDARY OUTCOMES:
Change From Baseline in MMDs | Baseline up to Week 12 (Weeks 1-12)
Percentage of Participants With ≥50% Reduction From Baseline in MMDs | Baseline up to Week 12 (Weeks 1-12)
Percentage of Participants With ≥75% Reduction From Baseline in MMDs | Baseline up to Week 12 (Weeks 1-12)
Change from Baseline in the Number of Monthly Headache Days | Baseline up to Week 12 (Weeks 1-12)
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 20
Number of Participants with Anti-drug Antibodies (ADA) | Up to Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (120):
- United States (28):
  - Accel Research Sites Network - Neurology and Neurodiagnostic of Alabama, Hoover, Alabama
  - Profound Research - Neurology Center of Southern California, Carlsbad, California
  - Neurology Center of North Orange County, Fullerton, California
  - CenExel CNS, Los Alamitos, California
  - ASCLEPES Research Centers, Sherman Oaks, California
  - Ki Health Partners LLC DBA New England Institute for Clinical Research, Stamford, Connecticut
  - K2 Medical Research - Winter Garden, Clermont, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - K2 Medical Research, LLC - Maitland, Maitland, Florida
  - Aqualane Clinical Research, Naples, Florida
  - K2 Medical Research Tampa LLC, Tampa, Florida
  - Premiere Research Institute Palm Beach, West Palm Beach, Florida
  - Accellacare and McFarland Clinic, Ames, Iowa
  - Clinical Research Professionals, Chesterfield, Missouri
  - Healthcare Research Network, Hazelwood, Missouri
  - Dent Neurosciences Research Center, Inc., Amherst, New York
  - North Suffolk Neurology, PC., Port Jefferson Station, New York
  - Accellacare of Cary - Cary Medical Group, Cary, North Carolina
  - Headache Wellness Center, Greensboro, North Carolina
  - Raleigh Medical Group, Raleigh, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Accellacare of Rocky Mount, Rocky Mount, North Carolina
  - Triad Neurological Associates, Winston-Salem, North Carolina
  - Accellacare of Charleston, Mt. Pleasant, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - Cedar Health Research, LLC, Dallas, Texas
  - Mercury Clinical Research, Sugar Land, Texas
  - MedStar Health - Neurology Clinic at McLean, McLean, Virginia
- Bulgaria (4):
  - Diagnostic Consultative Center Convex Ltd, Sofia, Sofiiska
  - MC Nevrocentrum, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sveti Georgi, Plovdiv
  - MC Rusemed-OOD, Rousse
- Czechia (11):
  - Neurosanatio s.r.o., Litomyšl, Pardubický kraj
  - Dr. Radomir Talab MD, Office of, Hradec Králové
  - Neuros s.r.o, Pilsen
  - Clintrial s. r. o., Prague
  - DADO MEDICAL s.r.o., Prague
  - Praglandia s.r.o, Prague
  - Axon Clinical s r.o, Prague
  - Neurologicka ordinace FORBELI sro, Prague
  - Institut neuropsychiatricke pece, Prague
  - Neurologicka ambulance, Slezská Ostrava
  - NeuroMed Zlin s.r.o., Zlín
- Denmark (2):
  - Bispebjerg Hospital - Region Capital, Copenhagen
  - Glostrup Hospital, Glostrup Municipality
- France (6):
  - Centre Hospitalier Universitaire de Lyon, Hopital Pierre Wertheimer, Bron
  - Centre Hospitalier Universitaire de Clermont Ferrand - Gabriel Montpied, Clermont-Ferrand Cedex1
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Roger Salengro, Lille
  - Assistance Publique Hopitaux de Marseille (AP-HM) - Hopital de La Timone, Marseille
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Lariboisiere, Paris
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital Pierre-Paul Riquet, Toulouse
- Georgia (8):
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
  - Caucasus Medical Center Ltd, Tbilisi
  - Archangel St Michael Multiprofile Clinical Hospital, Tbilisi
  - Jo Ann Medical Center, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Aversi Clinic, Tbilisi
  - MD Georgia Staff Physician MediClub Georgia, Tbilisi
  - S. Khechinashvili University Hospital, Tbilisi
- Germany (6):
  - Charite - Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - Studienzentrum Dr. Bischof GmbH, Böblingen
  - Klinik Haag i. OB, Ebersberg
  - Headache Center Frankfurt, Frankfurt
  - Siteworks - Hannover, Hanover
  - Siteworks - Heidelberg, Heidelberg
- Hungary (2):
  - S-Medicon Kft., Budapest, Central Hungary (Közép-Magyarország)
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Japan (16):
  - Jinnouchi Neurosurgery Clinic, Kasuga-shi, Fukuoka
  - Ikeda Neurosurgery Clinic, Kasuga-shi, Fukuoka
  - Nakamura Memorial Hospital, Sapporo, Hokkaid¿
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Tanaka Neurosurgery & Headache Clinic, Kagoshima, Kagoshima-ken
  - Atsuchi Neurosurgical Hospital, Kagoshima, Kagoshima-ken
  - Shonan Keiiku Hospital, Fujisawa-shi, Kanagawa
  - Sendai Headache and Neurology Clinic Medical Corporation, Sendai, Miyagi
  - Tominaga Hospital, Osaka, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Japanese Red Cross Shizuoka Hospital, Shizuoka, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-Gun, Tochigi
  - Shinagawa Strings Clinic, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Tokyo
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Klaipeda¿s University Hospital, Klaipėda
  - Medicum Centrum, Tauragė
  - Vilniaus Universiteto Medicinos Fakultetas - Neurologijos ir Neurochirurgijos Klinika - Neurologi..., Vilnius
- Poland (19):
  - Centrum Medyczne HCP sp. z o.o, Poznan, Greater Poland Voivodeship
  - Landa Specjalistyczne Gabinety Lekarskie, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Neuroprotect, Warsaw, Masovian Voivodeship
  - Neuro-Care sp. z o.o. sp. Komandytowa, Katowice, Silesian Voivodeship
  - Centrum Medczyne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzezicka Lekarze Spolka partnerska, Elblag
  - Pratia MCM Krakow, Krakow
  - Centrum Opieki Zdrowotnej OrkanMed, Ksawerów
  - Appletreeclinics Network Sp. z o.o., Lodz
  - Clinirem Sp. z o.o., Lublin
  - Indywidualna Praktyka Lekarska Dr hab. n. med. Anna Szczepanska-Szerej, Lublin
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin
  - Twoja Przychodnia NCM, Nowa Sól
  - Instytut Zdrowia dr Boczarska-Jedynak, Oświęcim
  - Neurologiczny Niepubliczny ZOZ Centrum Leczenia SM Osrodek Badan Klinicznych im. dr n. med. Hanki..., Plewiska
  - RCMed Oddzial Sochaczew, Sochaczew
  - MTZ Clinical Research Powered by Pratia, Warsaw
  - MIGRE Polskie Centrum Leczenia Migreny, Wroclaw
  - ClinHouse Centrum Medyczne, Zabrze
- Romania (3):
  - Sc Clubul Sanatatii S.R.L., Campulung Muscel, Judet Arges
  - Policlinica CCBR S.R.L., Bucharest
  - The Emergency County Clinical Hospital St. Andrew Constanta, Constanța
- Slovakia (4):
  - Private Practice - Dr. Beáta Dupejová, Banská Bystrica
  - IN MEDIC s.r.o, Bardejov
  - KONZILIUM s.r.o., Dubnica nad Váhom
  - SANERA, s.r.o., Prešov
- Spain (7):
  - Hospital General Universitario de Alicante, Alicante
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia (Instituto de Investigacion Sanitaria INCLIVA), Valencia
  - Hospital Universitario La Fe de Valencia, Valencia